CLINICAL TRIAL: NCT02645708
Title: External Physical Vibration Lithecbole(EPVL) Contrast With the Traditional Row of Stone Effect After Retrograde Intrarenal Surgery(RIRS): A Multi-center Prospective Randomized Controlled Trial
Brief Title: External Physical Vibration Lithecbole(EPVL) Versus Traditional Row of Stone After Retrograde Intrarenal Surgery(RIRS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice President of the Hospital, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRER(54)2015
Record Dates: First submitted 2015-12-07; First posted 2016-01-05 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-08

CONDITIONS: Renal Calculi
Keywords: RIRS; EPVL; PDI(Percussion,Diuresis,Inversion); Randomized Controlled Trial
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retrograde Intrarenal Surgery (RIRS) (Other): Patients in Group 1 undergo Retrograde Intrarenal Surgery
  Interventions: Procedure: Retrograde Intrarenal Surgery
- EPVL after RIRS (Other): Patients in Group 2 undergo external physical vibration lithecbole after Retrograde Intrarenal Surgery.
  with the help of changing the position and direction of the extracorporeally physical vibration machine, the urinary stone was discharged from the urinary collecting system
  Interventions: Procedure: EPVL after RIRS

INTERVENTIONS:
Procedure: Retrograde Intrarenal Surgery — Patients undergo Retrograde Intrarenal Surgery
  Arms: Retrograde Intrarenal Surgery (RIRS)
Procedure: EPVL after RIRS — Patients in Group 2 undergo EPVL after RIRS
  Arms: EPVL after RIRS

SUMMARY:
The treatment of renal calculus by retrograde intrarenal surgery(RIRS) isn't able to eliminate stone completely, hastening fragments clearance just only rely on traditional expulsive methods such as high fluid intake ,increasing physical activity, medical expulsive therapy and changing body position. Therefore, researchers purpose to evaluate the effectiveness of external physical vibration lithecbole(EPVL) in treatment of residual fragments after RIRS by prospective study of clinical trial, which will improve stone-free rate of residual fragments and benefit more patients.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of external physical vibration lithecbole for the treatment of residual stone after the operation of RIRS，thereby improving stone clearance rate. Investigators will do a multi-centers randomized controlled trial(RCT)，and investigators plan to perform this study in 10 hospitals，which are the First Affiliated Hospital of Guangzhou Medical University of China, Department of Urology, The Second Affiliated Hospital of Zhengzhou University of China, Jiangsu Province Hospital, Hubei Province Hospital, Zhongshan Hospital, Tongji Hospital,Hubei provincial people's Hospital,Guilin 181 Hospital，the People' Hospital of Huzhou，The People' Hospital of Shaoyang.

Investigators plan to beginning their study August 2015 and end July 2016. One hundred and eighty patients with postoperative residual stone after RIRS will be enrolled in this study. By simple random sampling technique, all the patients will be assigned to the segment of natural stone row group or physical row of stone group, compared two groups of patients with stone clearance rate and complications, Investigators hope that through this test, improve stone clearance rate after RIRS.

The principle of extracorporeal physical vibration:

A Simple harmonic motion technology in multi-direction was applied. The Lateral acceleration was provided by the physical vibration device in the base through the harmonic vibration wave in the horizontal direction, which induces the urinary stone separate with the kidney or ureter, and expands a moving space for the stone. Meanwhile, an axial effect was produced to push the stone by the physical vibration device in the handle through the harmonic vibration wave in the multi- direction. Finally, with the help of changing the position and direction of the extracorporeally physical vibration machine, the urinary stone was discharged from the urinary collecting system.

Number:

180cases(90 cases in control group, 90 cases in EPVL group)

Grouping methods:

In this trial, investigators use equilibrium randomization methods that generate random numerical code table, according to the table, patients are randomly assigned to different groups.

Evaluating indicator Stone-free rate in 5 weeks after RIRS. Incidence rate of complications and adverse reactions after EPVL(fever, hematuria).

Trial method; Cases selection and grouping: in 1 week after RIRS, the imaging KUB(abdominal plain film), patients with radiolucent calculus need to be examined by CT demonstrate the presence of residual fragments, and the cases that meeting inclusion criterion are randomly assigned to groups, and the ureteral stent should be removed in 2 weeks;

Laboratory testing: blood routine, urine routine, renal function , coagulation function; Strat the treatment of EPVL before the removal of ureteral stent.

Methods of control group(group1):

RIRS without EPVL Patients should be reexamined respectively in 1 and 2 weeks after RIRS, and the ureteral stent should be removed in 2 weeks;

Patients should follow the measures below:

1. the amount of fluid intake is more than 2000ml/d
2. increase physical activity
3. rest in position on uninjured side, patients with lower renal calyx calculus need to invert body;

Follow up timing: respectively in 2 ,3 and 5 weeks after RIRS.

Methods of EPVL group(group2):

Preparation before EPVL: the amount of fluid intake is about 1000-2000ml, start the treatment of EPVL when patient's bladder is filling;

Record: patients' information, outcome of treatment (examined by KUB right after EPVL); Start the treatment of EPVL;

Patients should follow the measures below:

1. the amount of fluid intake is more than 2000ml/d
2. increase physical activity
3. rest in position on uninjured side, patients with lower renal calyx calculus need to invert body;

Patients should be reexamined in one week, meanwhile removing ureteral stent or perhaps undergoing the treatment of EPVL once again.

Follow up timing: respectively in 1,2 and 4 weeks after EPVL..

Follow up project Laboratory testing: routine urinalysis; Imaging examination: KUB or kidney CT scan (radiolucent calculus) Complications and adverse reactions. Data gathering Fill in follow up table data; Radiological images; IVP(intravenous pyelography) or kidney CT scan; Reexamined by KUB (radiopaque calculus) or CT (radiolucent calculus) right after RIRS, respectively in 2 ,3 and 5 weeks after RIRS. If stones have been eliminated completely in patients with radiolucent calculus before or at the fourth week of follow-up, investigator must provide kidney CT scan.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-65 years;
2. The imaging demonstrate the presence of residual fragments in 1 week after RIRS;
3. Renal or upper ureteral calculus;
4. There's no urinary tract obstruction below stones, and stones didn't cause complete urinary tract obstruction;
5. Stones are fragmented successfully on single session of RIRS, and the diameter of any of fragments is less than 4mm;
6. Normal renal function.

Exclusion Criteria:

1. Couldn't tolerate EPVL;
2. Urinary tract anomalies, stricture or obstruction;
3. Calculus in diverticulum;
4. Severe hydronephrosis;
5. Combined with acute urinary tract infection;
6. Coagulation abnormalities;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change from stone free rate(SFR) with different follow-up periods | return hospital respectively in 2,3 and 5 week after RIRS
  Primary SFR is assessed by abdominal plain film （KUB）at2,3,5 week after operation. Stone-free status are defined as either the absence of any residual stone fragments.

SECONDARY OUTCOMES:
extracorporeal physical vibration complications | return hospital respectively in 2 ,3 and 5 weeks after RIRS
  Complication is defined as any adverse event occurred

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided